CLINICAL TRIAL: NCT02886390
Title: Intravenous Rt-PA Thrombolysis Combined With Remote Ischemic Post-Conditioning for Acute Ischemic Stroke Patients
Brief Title: r-tPA Thrombolytic Therapy in Combination With Remote Ischemic Conditioning for Acute Ischemic Stroke Recovery
Acronym: rtPA-RIC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Ji Xunming,MD,PhD, professor, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RIC-2016
Record Dates: First submitted 2016-08-28; First posted 2016-09-01 (Estimated); Last update posted 2018-06-20 (Actual); Status verified 2018-06

CONDITIONS: Stroke, Acute
Keywords: remote ischemic conditioning; r-tPA thrombolytic therapy
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RIC group (Experimental): The upper limb ischemic conditioning is composed of five cycles of bilateral upper limb ischemia intervened by reperfusion, which is induced by two cuff placed around the upper arms respectively and inflated to 200 mm Hg for 5 minutes followed by 5 minutes of reperfusion by cuff deflation. This therapy started within 2 hours after r-tPA thrombolytic therapy. In addition, all participants receive a standard clinical therapy.
  Interventions: Device: ischemic conditioning
- Control group (No Intervention): The participants received r-tPA thrombolytic therapy after diagnosed ischemic stroke. In addition, all participants receive a standard clinical therapy.

INTERVENTIONS:
Device: ischemic conditioning — In this study, the remote ischemic conditioning treatment was composed of five cycles of bilateral upper limb ischemia intervened by reperfusion, which was induced by two cuff placed around the upper arms respectively and inflated to 200 mm Hg for 5 minutes followed by 5 minutes of reperfusion by cuff deflation.
  Other Names: Doctormate, IPC-906
  Arms: RIC group

SUMMARY:
to detect the efficiency and safety of intravenous rtPA combined with RIPC in acute ischemic stroke patients

DETAILED DESCRIPTION:
Remote ischemic post-conditioning, which consists of several brief cycles of intermittent ischemia-reperfusion of the arm or leg, may potentially confer a powerful systemic protection against prolonged ischemia in a distant organ. Numerous reports have confirmed it strongest endogenous neuroprotection against brain injury after stroke. Ren et al demonstrated that remote ischemic post-conditioning (RIPC) performed in the hind limbs can not only significantly reduce the stroke volume within 3 hours in rat model, but also ameliorate the outcome of the behavioral test. A long-term repeated RIPC therapy can also help improving neurological functions. A combination of RIPC and tPA can help with neuroprotection which improves the neurological functions. Thus, it is meaningful to transform these basic experimental results to the clinical treatment. In the RECAST-1 trial, RIC has shown it safety and efficiency in AIS patients without tPA. However, there is no further explanation for the patients with IVT. Thus, in this study, we aim to demonstrate the efficiency and safety of RIPC in AIS patients performed rt-PA within 4.5 hours.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age≥18;
* Clinical sign and symptoms consistent with the diagnosis of an acute ischemic stroke, onset of stroke symptoms within 4.5 h before initiation of intravenous rt-PA thrombolytic therapy;
* Baseline National Institutes of Health Stroke Scale (NIHSS) score of 4-15 (assessed before intravenous alteplase), mRS ≤1 before onset of stroke symptom;
* No contraindication for MRI.
* Informed consent obtained

Exclusion Criteria:

* Cardioembolism；
* Contraindication for remote ischemic conditioning: severe soft tissue injury, fracture, or peripheral vascular disease in the upper limbs;
* Life expectancy < 1 year;
* Pregnant or breast-feeding women;
* Unwilling to be followed up or poor compliance for treatment; (5) Patients being enrolled or having been enrolled in other clinical trial within 3 months prior to this clinical trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-06-16 (Actual); Primary Completion 2019-02 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
infarction volume in brain between two groups | measured during 72 h
  assess by MRI-DWI and ADC

SECONDARY OUTCOMES:
The score of Modified Rankin scale score | measured at baseline(before RIPC),24 hours, at 5-7 days,30±7 days, 90±7 days
  The Modified Rankin Scale Score (mRS) is the most comprehensive and most widely used primary outcome measurement to assess the neurological functional disability in contemporary acute stroke trials. The mRS is an ordinal, graded interval scale that assigns patients among 7 global disability levels, which ranges from 0 (no symptom) to 5 (severe disability) and 6 (death). We will use mRS to evaluate the degree of disability or dependence during daily activities. The mRS will be assessed by certified study investigator, who is blinded to the treatment assignment, at 90 days postoperation. The distribution of mRS will be compared between groups
proportional of Modified Rankin scale scored 0-1 | measured at baseline(before RIPC),24 hours, at 5-7 days,30±7 days, 90±7 days
  The Modified Rankin Scale Score (mRS) is the most comprehensive and most widely used primary outcome measurement to assess the neurological functional disability in contemporary acute stroke trials. The mRS is an ordinal, graded interval scale that assigns patients among 7 global disability levels, which ranges from 0 (no symptom) to 5 (severe disability) and 6 (death). We will use mRS to evaluate the degree of disability or dependence during daily activities. The mRS will be assessed by certified study investigator, who is blinded to the treatment assignment, at 90 days postoperation. The distribution of mRS will be compared between groups
The score of National Institute of Health stroke scale score | measured at baseline(before RIPC),24 hours, at 5-7 days,30±7 days, 90±7 days
  National Institute of Health Stroke Scale (NIHSS) is considered as a standardized assessment of neurological functions in the acute phase of stroke, and it is generally used to quantify patient's neurological impairments on 15 items in 11 fields of different neurological status.The score of the scale ranges from 0 to 42.And higher score indicates worse neurological function.
The score of Barthel Index(BI) | measured at baseline(before RIPC),24 hours, at 5-7 days,30±7 days, 90±7 days
  the BI is used to measure performance in activities of daily living.The score of the scale ranges from 0 to 100. And lower score indicates worse activities of daily living.
recurrence of stroke and TIA | changes from baseline(before RIPC) to 90±7 days
  Stroke recurrence was defined as sudden functional deterioration in neurologic status with a decrease of 4 or more in the NIHSS, or a new stroke lesion on MRI/DWI located at the territory of the affected intracranial arteries.
death and any other adverse events | changes from baseline(before RIPC) to 90±7 days
  The investigator will record the number.
any ICH | changes from baseline(before RIPC) to 90±7 days
  Head computed tomography or magnetic reasoning imaging (MRI) scan will be performed to confirm intracerebral hemorrhage, and the imaging will be evaluated by two independent neuroradiologists who are blinded to the study assignment.
Distal radial pulses | during 90 days
  professional doctors will check the distal radial pulses
Visual inspection for local edema | during 90 days
  Professional oculists will check the fundus oculi to evaluate whether there is local edema.
The number of patients with erythema,and/or skin lesions related to RIC | during 90 days
  Professional doctors will check it and the investigator will record the number.
Palpation for tenderness | during 90 days
  Professional doctors will check it.
The number of patients not tolerating RIC procedure,and refuse to continue the RIC procedure | during 90 days
  The investigator will record the number.
the score of Numeric Rating Scale (NRS) | during 90 days
  The Numeric Rating Scale (NRS-11) is an 11-point scale for patient self-reporting of pain. The score from 0-10. the higher
the score of Hamilton Rating Scale for Depression（HAMAD） | change from baseline(before rtPA) to 90 days
  this score was used to provide an indication of depression, and as a guide to evaluate recovery.
level of MMP-9 | measured at baseline(before RIPC,after rtPA) and 7 days
  Blood samples will be drawn from cubital vein to test these biomarkers.These samples will be centrifuged immediately after collection and stored at - 80 until batch evaluation
level of IL-6 | measured at baseline(before RIPC,after rtPA) and 7 days
  Blood samples will be drawn from cubital vein to test these biomarkers.These samples will be centrifuged immediately after collection and stored at - 80 until batch evaluation
level of HS-CRP | measured at baseline(before RIPC,after rtPA) and 7 days
  Blood samples will be drawn from cubital vein to test these biomarkers.These samples will be centrifuged immediately after collection and stored at - 80 until batch evaluation
The level of vascular endothelial growth factor | measured at baseline(before RIPC,after rtPA) and 7 days
  Blood samples will be drawn from cubital vein to test these biomarkersThese samples will be centrifuged immediately after collection and stored at - 80 until batch evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Xunming Ji, MD. PhD, Principal Investigator — Xuanwu Hospital, Beijing
Locations (2):
- China (2):
  - Xuanwu Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Lu He hospital, Capital Medical University, Beijing, Beijing Municipality